CLINICAL TRIAL: NCT01769963
Title: Advanced Glycation End-products, Inflammation and Vascular Health in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: F111220003
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease
Keywords: Advanced glycation end-products; chronic kidney disease; nutrition; inflammation; insulin resistance; endothelial function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary intervention (Experimental): All participants will be fed a high AGE diet followed by a low AGE diet (single arm study)
  Interventions: Other: Research diet

INTERVENTIONS:
Other: Research diet — Participants will be provided specially prepared meals to eat at home for three weeks. During the first week, participants will eat foods that have standard amounts of AGEs in them (this is called the control diet). During the second and third weeks, participants will eat the same foods, only they will be prepared in our kitchen in a way that limits the amount of AGEs in them (called the intervention diet).

SUMMARY:
The purpose of the study is to learn more about how advanced glycation end-products can affect insulin resistance, inflammation and blood vessel health in people with kidney disease.

DETAILED DESCRIPTION:
Advanced glycation end-products (AGEs) are compounds that form when sugars abnormally attach to proteins or lipids. High levels of AGEs in the blood may cause inflammation, problems with controlling blood sugar, and problems with the health of blood vessels. Many of the foods we commonly eat have high amounts of AGEs, which may increase AGEs in the blood of people with kidney disease. The amount of AGEs in foods can be lowered when prepared using special cooking techniques such as using moist heat or longer cooking times at lower temperatures. New research has shown that preparing food in this way can lower inflammation and improve blood vessel health in people with normal kidney function.

In this study, the investigators would like to examine the effect of lowering the AGE content of foods on inflammation, blood sugar control, and blood vessel health in individuals with mild to moderate chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate CKD (estimated glomerular filtration rate 15 - 59 ml/min/1.73m2).

Exclusion Criteria:

* Current or past use of anti-glycemic medications
* Fasting glucose > 126 mg/dl on screening visit or positive glucose on urine dipstick
* Nephrotic-range proteinuria (≥ 3.5 grams per day as assessed by a spot urine albumin to creatinine ratio obtained at the screening visit)
* Pregnancy or breast-feeding
* Clinical need for a specialized diet (low sodium, low potassium, etc.) or religious dietary restrictions.
* New or recent change (< 3 months) in dosage of medications known to affect vascular reactivity- angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta-blockers, calcium channel blockers, HMG-CoA reductase inhibitors, etc.
* Current smoking or recent (< 6 months) cessation of smoking.
* Poorly controlled hypertension (≥ 140 mm Hg systolic or 90 mm Hg diastolic), or prior history of malignant hypertensive episode (SBP > 200) off of blood pressure medications.
* Participants with rapidly advancing renal failure.
* Severe anemia, defined as a hemoglobin < 8 g/dL for men and < 6 g/dL for women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
N-epsilon-carboxymethyllysine (CML) | baseline, one week and three weeks
  Change in CML concentrations
Inflammatory biomarkers | baseline, one week and three weeks
  Change in interleukins 1, 6 and 10, c-reactive protein
Indices of insulin sensitivity | baseline, one week and three weeks
  Change in HOMA-IR
Flow-mediated dilation (FMD) | one week and three weeks
  Changes in brachial FMD

CONTACTS AND LOCATIONS:
Overall Officials: Orlando M Gutiérrez, MD, MMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States